CLINICAL TRIAL: NCT05688566
Title: 攀爬機踏板在不同角度下對於下肢生物力學影響 Biomechanical Characteristics of Lower Extremity During Pinnacle Trainer With Different Pedal Angles.
Brief Title: Biomechanical Characteristics of Lower Extremity During Pinnacle Trainer With Different Pedal Angles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Distinguished Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 111-356
Record Dates: First submitted 2022-12-25; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Healthy Adult
Keywords: biomechanical characteristics of lower extremity; Pinnacle trainer; pedal angles

STUDY DESIGN:
Intervention Model Description: Then the pedal angle are inversion 10 ˚,0 ˚, eversion 10˚. Participants stepped on the Pinnacle trainer under three angle levels, namely inversion 10 ˚,0 ˚, eversion 10˚.
Masking Description: The subject already knows the angle of the pedal when he steps on the pedal, because there are only three angles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- zero condition (Experimental): Then the pedal angle is the angle between the lowest pedal position and the floor. The zero condition is 0 ˚of pedal angle.Participants were asked to step with the consistent cadence at 60 steps/ min by the metronome.Three successful trials will be collected for each condition. Fifteen seconds of data will be collected for each trial.
  Interventions: Device: pinnacle trainer
- eversion codition (Active Comparator): Then the pedal angle is the angle between the lowest pedal position and the floor. The eversion condition is -10 ˚of pedal angle.Participants were asked to step with the consistent cadence at 60 steps/ min by the metronome.Three successful trials will be collected for each condition. Fifteen seconds of data will be collected for each trial.
  Interventions: Device: pinnacle trainer
- inversion condition (Active Comparator): Then the pedal angle is the angle between the lowest pedal position and the floor. The inversion condition is +10 ˚of pedal angle.Participants were asked to step with the consistent cadence at 60 steps/ min by the metronome.Three successful trials will be collected for each condition. Fifteen seconds of data will be collected for each trial.
  Interventions: Device: pinnacle trainer

INTERVENTIONS:
Device: pinnacle trainer — The pinnacle trainer (S776MA, SportsArt, Taiwan) was used in this study.

SUMMARY:
To investigate the effects of pedal degree on the biomechanical characteristics of the healthy adults' lower limbs during stepping on the pinnacle trainer.The purpose of this study are compare the biomechanical characteristics of low limbs at different angle of pedal during stepping on Pinnacle trainer. The investigators hope to provide this outcome to therapists can make the rehabilitation training more effective and delay the disease progression of KOA patients.

DETAILED DESCRIPTION:
The pedal angle influences the force distribution in the lower extremities. Although we have seen the angle of the pedal selected of the bicycle and a lot of insole paper, the previous paper did not see adjusting the pedal angle of the pinnacle trainer. However, the joint loading and force distribution during stepping on a pinnacle trainer with various pedal angle are unknown. The investigation of biomechanics of the lower extremity is important to provide information about the joint loadings and prevent potential injuries during exercise.According to the World Health Organization, by 2050, people over 60 years old will account for nearly 22% of the world's population. Of that 22%, a conservative estimate of 15% will have symptomatic OA. It is estimated that by 2050, nearly 130 million people worldwide will suffer from OA, and 40 million people will gradually affect their lives and be severely disabled due to osteoarthritis by 2050. Knee Osteoarthritis accounts for more than 80% of the global OA disease burden. And previous studies suggested that the use of the Pinnacle Trainer for individual with knee OA is effective on the improvement of pain intensity, physical functions and the muscular strength of the low extremity. And the internal knee abduction moment demonstrated a tendency toward to reduce after the Pinnacle Trainer intervention. Hence, the reduction of excessive internal knee abduction moment is beneficial for some users. On the other hand, the internal knee abduction moment is related to the severity of the knee OA.

The majority of research has focused specifically on the effect of lateral wedge insoles at the knee, and numerous of studies have concentrated on pedals on stationary cycling. Those studies suggested that the foot everted position reduced the KAM. However, few studies investigated the angle of pedal during the CKC exercise equipment. However, the biomechanical characteristics during stepping on Pinnacle Trainer with different pedal angles are unknown. The investigators wanted to explore the biomechanical characteristics of lower extremity during pinnacle trainer with different pedal angles and further explore whether KAM can be effectively reduced by changing the angle of the wedge to assist the training of KOA patients.

The purpose of this study are compare the biomechanical characteristics of low limbs at different angle of pedal during stepping on Pinnacle trainer. The investigators hope to provide this outcome to therapists can make the rehabilitation training more effective and delay the disease progression of KOA patients.

ELIGIBILITY:
Inclusion Criteria:

30 healthy individuals above 20 years and will be recruited in this study. 30 participants will be recruited with considering the inclusion criteria as follows:

1. 20 years old above
2. Able to perform regular exercise
3. Able to understand Chinese or Taiwanese language
4. Healthy adult (no skeletal muscle, neurological disease, normal BMI (18.5≦BMI<25.0), and no disease that will affect training.

Exclusion Criteria:

1. Having illness or diseases that cannot perform physical exercise
2. Having any kinds of chronic disease that might be more activated by performing Pinnacle training such as cardiovascular diseases, chronic respiratory diseases, osteoporosis, etc.
3. Having chronic diseases that cannot perform Pinnacle training according to the experimental protocols such as blindness, deafness and hearing impairment, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
lower limb movement | 2 hours
  A three-dimensional motion capture system with eight digital cameras (Osprey, Motion Analysis Corporation, USA) was used to collect the data of low limb motion. The sampling rate was set at 200 Hz. Reflective markers (10 mm in diameter) will be attached on the participant's skin at the positions with regards to Modified Helen-Hayes marker set.
kinetics of lower limb | 2 hours
  Two six-axis force and torque transducers (Mini85, ATI Industrial Automation, USA) with a sampling rate of 1000 Hz were placed under the pedals of the pinnacle trainer.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu TW, Chien HL, Chen HL. Joint loading in the lower extremities during elliptical exercise. Med Sci Sports Exerc. 2007 Sep;39(9):1651-8. doi: 10.1249/mss.0b013e3180dc9970. PMID 17805099
- [Background] You YL, Lin CJ, Chieh HF, Tsai YJ, Lee SY, Lin CF, Hsu YC, Kuo LC, Su FC. Comparison of knee biomechanical characteristics during exercise between pinnacle and step trainers. Gait Posture. 2020 Mar;77:201-206. doi: 10.1016/j.gaitpost.2020.02.003. Epub 2020 Feb 4. PMID 32058284
- [Background] Stauffer RN, Chao EY, Brewster RC. Force and motion analysis of the normal, diseased, and prosthetic ankle joint. Clin Orthop Relat Res. 1977;(127):189-96. PMID 912978
- [Background] Foroughi N, Smith R, Vanwanseele B. The association of external knee adduction moment with biomechanical variables in osteoarthritis: a systematic review. Knee. 2009 Oct;16(5):303-9. doi: 10.1016/j.knee.2008.12.007. Epub 2009 Mar 24. PMID 19321348
- [Background] Haim A, Wolf A, Rubin G, Genis Y, Khoury M, Rozen N. Effect of center of pressure modulation on knee adduction moment in medial compartment knee osteoarthritis. J Orthop Res. 2011 Nov;29(11):1668-74. doi: 10.1002/jor.21422. Epub 2011 Apr 13. PMID 21491477
- [Background] Chang SY, Lin YJ, Hsu WC, Hsieh LF, Lin YH, Chang CC, Chou YC, Chen LF. Exercise Alters Gait Pattern but Not Knee Load in Patients with Knee Osteoarthritis. Biomed Res Int. 2016;2016:7468937. doi: 10.1155/2016/7468937. Epub 2016 Sep 20. PMID 27725941
- [Background] Thorp LE, Wimmer MA, Foucher KC, Sumner DR, Shakoor N, Block JA. The biomechanical effects of focused muscle training on medial knee loads in OA of the knee: a pilot, proof of concept study. J Musculoskelet Neuronal Interact. 2010 Jun;10(2):166-73. PMID 20516634
- [Background] Butler RJ, Marchesi S, Royer T, Davis IS. The effect of a subject-specific amount of lateral wedge on knee mechanics in patients with medial knee osteoarthritis. J Orthop Res. 2007 Sep;25(9):1121-7. doi: 10.1002/jor.20423. PMID 17469197
- [Background] Hinman RS, Bowles KA, Metcalf BB, Wrigley TV, Bennell KL. Lateral wedge insoles for medial knee osteoarthritis: effects on lower limb frontal plane biomechanics. Clin Biomech (Bristol). 2012 Jan;27(1):27-33. doi: 10.1016/j.clinbiomech.2011.07.010. Epub 2011 Sep 8. PMID 21862189
- [Background] Kean CO, Bennell KL, Wrigley TV, Hinman RS. Modified walking shoes for knee osteoarthritis: Mechanisms for reductions in the knee adduction moment. J Biomech. 2013 Aug 9;46(12):2060-6. doi: 10.1016/j.jbiomech.2013.05.011. Epub 2013 Jun 14. PMID 23768609
- [Background] Resende RA, Kirkwood RN, Deluzio KJ, Hassan EA, Fonseca ST. Ipsilateral and contralateral foot pronation affect lower limb and trunk biomechanics of individuals with knee osteoarthritis during gait. Clin Biomech (Bristol). 2016 May;34:30-7. doi: 10.1016/j.clinbiomech.2016.03.005. Epub 2016 Mar 24. PMID 27060435
- [Background] Fisher DS, Dyrby CO, Mundermann A, Morag E, Andriacchi TP. In healthy subjects without knee osteoarthritis, the peak knee adduction moment influences the acute effect of shoe interventions designed to reduce medial compartment knee load. J Orthop Res. 2007 Apr;25(4):540-6. doi: 10.1002/jor.20157. PMID 17205556
- [Background] Gregersen CS, Hull ML, Hakansson NA. How changing the inversion/eversion foot angle affects the nondriving intersegmental knee moments and the relative activation of the vastii muscles in cycling. J Biomech Eng. 2006 Jun;128(3):391-8. doi: 10.1115/1.2193543. PMID 16706588
- [Background] Gardner JK, Klipple G, Stewart C, Asif I, Zhang S. Acute effects of lateral shoe wedges on joint biomechanics of patients with medial compartment knee osteoarthritis during stationary cycling. J Biomech. 2016 Sep 6;49(13):2817-2823. doi: 10.1016/j.jbiomech.2016.06.016. Epub 2016 Jun 23. PMID 27451059
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Zimmermann CL, Cook TM, Bravard MS, Hansen MM, Honomichl RT, Karns ST, Lammers MA, Steele SA, Yunker LK, Zebrowski RM. Effects of stair-stepping exercise direction and cadence on EMG activity of selected lower extremity muscle groups. J Orthop Sports Phys Ther. 1994 Mar;19(3):173-80. doi: 10.2519/jospt.1994.19.3.173. PMID 8156070